CLINICAL TRIAL: NCT05093868
Title: Electrographic Flow Mapping VALidation in Patients With Persistent Atrial Fibrillation (EVAL AF)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Required equipment could not be obtained
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-021
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation
Keywords: electrographic flow mapping; EGF; atrial fibrillation; FIRMap; Abbott Laboratories; EGF Maps; HD Grid Maps
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FIRMap™ (Abbott Laboratories, Abbott Park, IL) (Experimental): A 64-pole basket mapping catheter (FIRMap™, Abbott Laboratories, Abbott Park, IL) will be used to passively acquire electrical signals
  Interventions: Device: Electrographic Flow Mapping

INTERVENTIONS:
Device: Electrographic Flow Mapping — Electrographic Flow Mapping will be collected

SUMMARY:
This is a prospective, observational, single center pilot trial to find out if a new computerized technology for analysis of the electrical activity recorded during atrial fibrillation can identify the electrical source of this arrhythmia. If we are able to reliably identify the source, then in the future we may be able to use this technology to determine the optimal sites for catheter ablation of atrial fibrillation in the heart. The present study will compare the standard electrical recordings to the new computerized algorithm analysis of recordings gathered at the same time. The study will enroll 30 participants with persistent or longstanding persistent atrial fibrillation (AF) that are scheduled for elective catheter ablation of AF. The catheters that are being placed in the heart are standard Food and Drug Administration (FDA)-approved mapping catheters. The investigational computerized software that will be employed in the trial will be used after the case has done and will not directly impact any of the activities during the ablation procedure. Information learned from this trial will improve understanding of the mechanisms of atrial fibrillation and will potentially improve success rates of AF ablation for patients in the future and will be used to design a prospective trial.

DETAILED DESCRIPTION:
It is hypothesized that initiation and propagation of atrial fibrillation (AF) is dependent, at least in part, on rapid atrial stimulation from focal sources. It is debated whether the mechanism of arrhythmogenesis at these foci is abnormal automaticity, triggered activity, microreentry or rotational reentry. However, after activation emerges from these "driver" sites, fibrillatory conduction ensues resulting in the disorganized conduction pattern of AF. Conventional mapping systems can either achieve high spatial resolution by sequential tachycardia beats following a fixed intra-atrial activation pattern (as in macro reentrant atrial flutter), or high temporal resolution with very low spatial resolution achieved through multielectrode basket catheters. Activation mapping in AF with commercially available mapping systems has been unsuccessful in identifying driver sites because atrial activation patterns change on a beat-to-beat basis precluding the use of sequential mapping approaches, and real-time mapping with basket electrodes lacks sufficient resolution to delineate the complex patterns of conduction. Electrographic Flow (EGF) mapping (AblaMap®, Ablacon, Inc, Wheat Ridge, CO) is a unique method to assess dominant patterns of intra-atrial conduction during ongoing atrial fibrillation and has been previously described. Recordings from a multielectrode basket catheter are analyzed for electrical activation vectors over sequential 2-second segments during a 60 second acquisition period. Patterns of reproducible vector activation are used to identify driver sources for the AF. Multiple sources are often identified in patients with persistent AF. It is anticipated that substrate modification of these source regions will eliminate the AF drivers and result in a favorable response to catheter ablation.

Participants undergoing elective catheter ablation of AF will be enrolled. During the elective catheter ablation and during ongoing AF, A 64-pole basket mapping catheter (FIRMap™, Abbott Laboratories, Abbott Park, IL) will be inserted into the right atrium, and electrical signals will be passively acquired. This is the only aspect of the procedure that will be research beyond standard of care. A 16-pole HD grid mapping catheter (Advisor™ HD Grid, Abbott Laboratories, Abbott Park, IL) will be inserted into the right atrium and high density electrogram signals will be recorded from each site for 2 minutes. At least 6 sites will be assessed. After transseptal catheterization, mapping of the left atrium will proceed in a similar fashion. Electrogram signals will be recorded in the electroanatomical mapping system as well as the 128-channel electrophysiology recording system. The collected electrogram data will be analyzed post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective catheter ablation of AF
* History of persistent or longstanding persistent AF (see definitions below)
* Able to provide written informed consent prior to the procedure
* Age ≥18 years

Exclusion Criteria:

* Ineligible to undergo elective atrial fibrillation ablation procedure due to medical illness or poor medical condition
* Presence of a permanent endocardial pacemaker or ICD (implantable cardioverter defibrillator)
* Presence of a prosthetic mitral heart valve
* Known reversible causes of AF including clinical hyperthyroidism, pericarditis/pleuritis or other active systemic inflammatory disease including post pericardiotomy syndrome, systemic lupus erythematosus, sarcoidosis and rheumatoid arthritis
* Decompensated clinical heart failure (NYHA class 4)
* Any cerebral ischemic event (strokes or transient ischemic attacks) which occurred during the 6-month interval preceding the consent date
* History of systemic thromboembolic event defined as clinical and arteriographic evidence of thromboembolism to any distal arterial vascular bed within the past 6 months, or evidence of intracardiac thrombus at the time of the procedure
* Pregnancy (pre-procedure pregnancy serum test will be performed in all premenopausal women)
* Unable to provide own informed consent due to cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-02 (Estimated); Primary Completion 2022-09-02 (Estimated); Study Completion 2022-09-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with correlation in detection of sources of atrial fibrillation between the electrographic flow (EGF) mapping multielectrode basket catheter and the high-density (HD) regional mapping catheter. | During elective catheter ablation procedure, an average duration of 3 to 6 hours
  The number of participants will be reported who have the same areas identified for primary sources of AF, secondary sources of AF and passive flow regions, using the two catheter modalities.

SECONDARY OUTCOMES:
AF cycle length calculated from EGF mapping catheter | Two-minute time intervals during elective catheter ablation procedure, an average duration of 3-6 hours
  Calculated mean AF cycle length in milliseconds as recorded using the EGF mapping multielectrode basket catheter
AF cycle length calculated from HD grid regional mapping catheter | Two-minute time intervals during elective catheter ablation procedure, an average duration of 3-6 hours
  Calculated mean AF cycle length in milliseconds as recorded using the HD grid regional mapping catheter

CONTACTS AND LOCATIONS:
Overall Officials: Nishaki Mehta, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No